CLINICAL TRIAL: NCT04850755
Title: A Phase I Dose Escalation Study of Selinexor Plus Nivolumab and Ipilimumab in Advanced/Metastatic Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7EL (BMS); IST-313 (KPT)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advance Solid Malignancies; Metastatic Solid Malignancies
Keywords: selinexor; nivolumab; ipilimumab
MeSH Terms: interventions — selinexor; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: For all patients, the phase I drug combination will be preceded by a 14-day run in period where selinexor alone will be administered and biopsies will be obtained both pre-and post selinexor dosing. Patients will be treated with all three drugs until disease progression (as defined by RECIST criteria) or intolerable drug toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with advanced solid malignancies (Experimental): Patients will be dosed with selinexor once a week continuously in a 6 week cycle. Nivolumab will be administered on biweekly of each cycle . Ipilimumab will be dosed only on D1 of each cycle . Ipilimumab will continue for a maximum of 4 cycles. Nivolumab and selinexor will continue for up to 24 months or until discontinuation criteria is met.
  Interventions: Drug: Selinexor in combination with nivolumab and ipilimumab

INTERVENTIONS:
Drug: Selinexor in combination with nivolumab and ipilimumab — Patients will commence at dose level 1. One cycle is 42 days (6 weeks) for all three agents. At dose level 1, selinexor will be dosedorally weekly, and nivolumab at 2 weekly + ipilimumab 1mg/kg 6 weekly. Patients can have dosing interruptions or reductions of any drug independently of one another, depending on the drug causing the toxicity

SUMMARY:
This is a single-centre, phase 1a (dose escalation) and 1b (dose expansion) study to evaluate the safety and tolerability of oral Selinexor in combination with nivolumab and ipilimumab in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the safety and tolerability of selinexor in combination with nivolumab and ipilimumab
* To determine the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended phase 2 dose (RP2D) of selinexor in combination with nivolumab and ipilimumab in patients with advanced or metastatic solid tumor malignancies.

Secondary Objectives

* To determine Selinexor pharmacokinetics (PK) in Asian patients
* To describe anti-tumor responses with the combination in patients with advanced or metastatic solid tumor malignancies.

Exploratory Objectives

* To assess the immunomodulatory effects of selinexor in solid tumour malignancies and circulating immune cells
* To identify biomarkers of response to the combination of selinexor and nivolumab + ipilimumab. We will explore changes in PDL1 expression, T cell infiltration (including CD4 and CD8 positive cells), gene expression profiles on serial tumor biopsies pre-selinexor, post-selinexor alone, and after the combination of selinexor and ipilimumab + nivolumab where feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. Willing and able to provide written informed consent in accordance with local institutional guidelines.
3. Dose Escalation Phase: Patients with histologically or cytologically confirmed advanced or metastatic solid tumors who have radiological evidence of progressive disease on study entry that is deemed unlikely to benefit from further standard therapy.
4. Dose Expansion phase: Patients with previously treated, metastatic or advanced recurrence malignancy confirmed histologically or cytologically. Patients must have evidence of progressive disease on study entry that is deemed unlikely to benefit from further standard therapy.
5. There is no upper limit on the number of prior treatments. Hormone ablation therapy is considered an anticancer regimen. Radiation and surgery are not considered anticancer regimens.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1.
7. Adequate hepatic function within 14 days prior to C1D1:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to <3 × ULN.
8. Adequate renal function within 14 days prior to C1D1 as determined by serum creatinine of ≤1.5 mg/dL OR estimated creatinine clearance of ≥ 30 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female.
9. Adequate hematopoietic function within 14 days prior to C1D1. Transfusions and growth factors are allowed prior to and throughout the study.

   1. Total white blood cell (WBC) count ≥1500/mm3, absolute neutrophil count ≥1000/mm3
   2. Hemoglobin ≥9 g/dL
   3. Platelet count ≥125,000/mm3 in dose escalation phase, and platelet count ≥100,000/mm3 in dose expansion phase.
10. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 5 months following the last dose of study treatment.

    a. Female patients of childbearing potential and fertile male patients must agree to use highly effective contraception listed below (ie, results in a low failure rate when used consistently and correctly) during the dosing period and for a period of at least 5 months after the end of treatment.

    b. Highly effective methods include: i. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

1. oral 2. intravaginal 3. transdermal ii. progestogen-only hormonal contraception associated with inhibition of ovulation:

1. oral
2. injectable
3. implantable iii. intrauterine device iv. intrauterine hormone-releasing system v. bilateral tubal occlusion vi. vasectomized partner vii. sexual abstinence

Exclusion Criteria:

Exclusion criteria 1. Patients with significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; 2. Radiation (except planned or ongoing palliative radiation to bone outside of the region of measurable disease) ≤ 3 weeks prior to cycle 1 day 1 3. Chemotherapy, or immunotherapy or any other systemic anticancer therapy ≤ 3 weeks prior to cycle 1 day 1.

4. Uncontrolled active infection requiring systemic antibiotics (Hepatitis B and C infection are NOT exclusion criteria).

1. Subjects with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/ml prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed. Subjects with Human Immunodeficiency Virus (HIV) who have CD4+ T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections in the last year are allowed.

5. Major surgery within 2 weeks of first dose of study drug. 6. Patients who are pregnant or breast-feeding; 7. Patients with significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications.

8. Patients with serious psychiatric or medical conditions that could interfere with treatment.

9. History of organ allograft 10. Patients who had previous grade 4 immune related adverse events from prior immunotherapy (including anti PD-1/PD-L1 or anti CTLA-4 antibodies).

11. Patients who previously received Selinexor and had grade 4 non laboratory adverse events that were considered treatment related or possibly treatment related.

12. Concurrent therapy with approved or investigational anticancer therapeutics; 13. Patients receiving chronic treatment with systemic steroid therapy (>10 mg/day prednisone or equivalent) within 7 days of the first dose of study treatment, other than replacement-dose steroids in the setting of adrenal insufficiency. Topical,inhaled, nasal and ophthalmic steroids are not prohibited.

14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

1. Subjects with vitiligo or alopecia
2. Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
3. Any chronic skin condition that does not require systemic therapy
4. Subjects without active disease in the last 5 years may be included but only after consultation with the medical monitor
5. Subjects with celiac disease controlled by diet alone
6. For other autoimmune or inflammatory conditions not specifically mentioned - to discuss on case by case basis with investigator and medical monitor 15. BSA <1.35 m2 (BSA calculated by Dubois or Mosteller methods)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Objective disease response assessment | 3 years
  to be made according to standard, international RECIST 1.1 criteria for solid tumors.
progression free survival (PFS) | 3 years
  the time interval from the starting date of combination treatment to the date of disease progression on treatment
duration of response (DOR) | 3 years
  is defined as the time from documentation of tumor response to disease progression
Duration of stable disease | 3 years
  is defined as the time from first RECIST assessment scan documenting stable disease by RECIST criteria, to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: David Shao Peng Tan, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galon J, Bruni D. Approaches to treat immune hot, altered and cold tumours with combination immunotherapies. Nat Rev Drug Discov. 2019 Mar;18(3):197-218. doi: 10.1038/s41573-018-0007-y. PMID 30610226
- [Background] Tan DS, Bedard PL, Kuruvilla J, Siu LL, Razak AR. Promising SINEs for embargoing nuclear-cytoplasmic export as an anticancer strategy. Cancer Discov. 2014 May;4(5):527-37. doi: 10.1158/2159-8290.CD-13-1005. Epub 2014 Apr 17. PMID 24743138
- [Derived] R Choo J, Jeraj SN, Sundar R, Yong WP, Lee M, Huang Y, Asokumaran Y, Chan GHJ, Ngoi NYL, Wong ALA, Soo RA, Chee CE, Lim JSJ, Goh BC, Lee SC, Tan DSP. NEXUS: a phase I dose escalation study of selinexor plus nivolumab and ipilimumab in Asian patients with advanced/metastatic solid malignancies. Ther Adv Med Oncol. 2025 Jun 9;17:17588359251339930. doi: 10.1177/17588359251339930. eCollection 2025. PMID 40502306